CLINICAL TRIAL: NCT01392820
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of TC-5214 in Japanese Healthy Elderly Male and Female Volunteers
Brief Title: A Study of Single and Multiple Ascending Doses of TC-5214 in Japanese Healthy Elderly Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D4131C00003
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Phase I; Japan; Elderly; PK; SAD; MAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-5214 (Experimental)
  Interventions: Drug: TC-5214
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Tablet, Oral, twice daily
  Arms: TC-5214
Drug: Placebo — Tablet, Oral, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, tolerability and pharmacokinetics of TC-5214 in elderly healthy Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy elderly male and female ≥65 years old.
* Have a BMI of ≥18 and ≤27 kg/m2 and weigh ≥ 45 kg.
* Be able to understand and comply with the requirements of the study as judged by the investigator(s).

Exclusion Criteria:

* History of any clinically significant medical or neurologic disease or disorder.
* History of gastrointestinal surgery or unintentional rapid weight loss.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the study drug.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
assess the safety and tolerability during single and multiple ascending oral doses by assessment of AEs, brief neurological examinations, vital signs, eye symptoms question, physical examinations, laboratory parameters, and ECGs, and C-SSRS. | During the whole study period, ca. 50 days

SECONDARY OUTCOMES:
characterise the PK of TC-5214 in plasma and urine during single and multiple ascending oral doses to Japanese healthy elderly volunteers. | PK samplings are taken at defined timepoints during residential periods, 4 days for SAD part and/or 9 days for MAD part.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Eriksson, MD, Study Director — AstraZeneca; Shunji Matsuki, MD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Fukuoka, Japan

REFERENCES:
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516